CLINICAL TRIAL: NCT05809856
Title: A First-in-Human Feasibility Study to Evaluate the Safety (and Short Term Effectiveness) of the Autologous GrOwnValve Transcatheter Pulmonary Heart Valve [GECT]
Brief Title: Feasibility Study to Evaluate the Safety of the Autologous GrOwnValve Transcatheter Pulmonary Heart Valve
Acronym: GECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: GrOwnValve GmbH (Unknown)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Frank Edelmann, Univ.-Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100592731
Record Dates: First submitted 2022-12-05; First posted 2023-04-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Valve Insufficiency
Keywords: Heart Valve Replacement; Pulmonary Valve; Congenital Heart Diseases; Transcatheter Valve; Medical Need; Durable; One-time-solution; Autologous Living Tissue
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Non-inferiority analysis with standard of current medical care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implantation of autologous GrOwnValve (Experimental): Implantation of autologous GrOwnValve via minimal-invasive transcatheter technique into patients with high-grade pulmonary valve insufficiency and right ventricular dilatation.
  Interventions: Device: GrOwnValve - novel heart valve replacement approach

INTERVENTIONS:
Device: GrOwnValve - novel heart valve replacement approach — The autologous GrOwnValve is implanted into a stent before it is implanted via minimal-invasive transcatheter technique into the patients with high-grade pulmonary valve insufficiency and right ventricular dilatation. Control intervention/Reference test: Since the study is designed for investigating the safety of the procedure, there will not be a control group. However, the outcomes will be compared as a non-inferiority analysis with the standard of current medical care (Edwards SAPIEN 3 or Medtronic's Melody, both bioprosthetic transcatheter pulmonary valves).

SUMMARY:
Aim of this study is to investigate the clinical safety of a novel pediatric heart valve.

DETAILED DESCRIPTION:
Defective or diseased pulmonary heart valves do not recover. If left untreated, pediatric and adult patients alike, face serious risks of progressive heart failure and death. Due to the insufficient care of children with heart valve defects, the valve replacement with regenerative, remodeling, and growth potential remains an unmet medical need. Therefore, the first pediatric heart valve (GrOwnValve) was developed to overcome the current limitations, which should offer regenerative potential that adapts to the somatic growth of the child. The study aims to investigate the safety and provide the first initial efficacy estimates of the transcatheter implantable GrOwnValve. This first prospective, non-randomized, single center trial in 7 study subjects (≥ 18 years of age) should be conducted to assess the devices safety for clinical application.

The novel interdisciplinary solution approach is based on the combination of individualized 3D modeling, viable autologous tissue (contrary to all other prosthetic heart valves on the market), and preservation of the regenerative capacity of the valve replacement by maintaining the vitality of heart valve cells and tissue through the application of a novel crosslinker in the tissue preparation process. The GrOwnValve prothesis has the potential to be the first durable and regenerative heart valve for adults. Fabrication is performed on-demand in the operating room. The trial should be the first clinical investigation assessing this novel heart valve replacement approach. We are aiming for the GrOwnValve to be the standard of care, replacing current solutions.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Sufficient appropriate tissue (preferably: Pericardium for pericardiectomy via thoracoscopy or thoracotomy, or sternotomy; other options are fascia lata, rectus fascia, peritoneum or diaphragm)
3. Any of the following by transthoracic echocardiography and/or Cardiac Magnet Resonance Imaging:

   * For patients in New York Heart Association (NYHA) Classification II, III, or IV: Moderate (3+) or severe (4+) pulmonary regurgitation AND/OR mean systolic gradient across PV or RVOT ≥ 35 mmHg
   * For patients in NYHA Classification I: Severe (4+) pulmonary regurgitation with RV dilatation or dysfunction and/or mean PV or RVOT systolic gradient ≥ 40 mmHg
   * Right ventricular ejection fraction (RV-EF): <40%.
   * Right ventricular end-diastolic volume (RVEDV): >150 ml/m2 (body surface area)
4. Written informed consent provided by study subjects obtained before any research-related test is performed

Exclusion Criteria:

* Active endocarditis or myocarditis or within 3 months before the screening date
* Patients unwilling or unable to provide written informed consent or comply with follow-up requirements
* Obstruction of the central veins (including the superior and inferior vena cava, and bilateral iliac veins) such that the Ensemble-delivery system/ Performer™ - Guiding Sheath/ Extra Large Check-Flo® or GORE® DrySeal Flex + Ballon-in-Ballon-catheter cannot be advanced to the heart via a transvenous approach from either femoral vein or internal jugular
* Requires emergency surgery
* Recipient of transplanted organs or currently an organ transplant candidate
* Pulmonary hypertension
* Connective tissue disorders
* Coronary artery disease
* Immunosuppressive disease
* Estimated survival of less than 6 months
* Fertile females unable to take adequate contraceptive precautions (PEARL- Index < 1%)
* Females who are pregnant, or are currently breastfeeding an infant
* Acute myocardial infarction within 30 days of the screening date
* Stroke confirmed by CT, cerebrovascular accident (CVA), or transient ischemic attack (TIA) within 6 months before the screening date
* Hemodynamic or respiratory instability requiring inotropic or/and mechanical circulatory support, or mechanical ventilation within 30 days before the screening date
* Severe left ventricular systolic dysfunction with ejection fraction ≤ 20% or evidence of an intra-cardiac mass, thrombus, or vegetation assessed by echocardiography before the screening date
* Renal insufficiency with creatinine level 2.5 mg/dl within 60 days before the screening date
* Leukopenia with WBC <3.5 x 109/L anemia with Hgb <10 g/dl, or thrombocytopenia with platelet count <50x103/l accompanied by a history of bleeding diathesis or coagulopathy within 60 days before the screening date
* Adult subject is an illicit drug user, alcohol abuser, or unable to give informed consent
* Subject is institutionalized by court order or by order of authority (e.g. prisoner, untreated psychiatry; limited compliance)
* Major or progressive non-cardiac disease (liver failure, renal failure, cancer)that has a life expectancy of less than six months Inability to comply with all of the study procedures and follow-up visits
* Subjects who are dependent on the sponsor or investigators

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2031-01-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | Up to 5 Years Follow-Up
  (valve-related, sudden, cardiac, and all-cause death)
Major bleeding | Up to 1 Year Follow-Up
  Assessment if device-related major bleeding has occured by laboratory + echo + CT
Reoperation | Up to 5 Years Follow-Up
  Questioning if device-related re-operation occured
Acute device-related complications | Up to 5 Years Follow-Up
  Measurement tool: Spiroergometry
  o Parameters: cardiac rhythm, load duration, reason for termination, Heart rate at rest, blood pressure, maximum load level, VE/VCO2, PetCO2, VE/VCO2 slope, VO2, Respiratory rate, VD/VT, SpO2, RER, Borg score, FEV1, FVC
Oxygen supply | Up to 5 Years Follow-Up
  Measurement tool: Spiroergometry Parameters: cardiac rhythm, load duration, reason for termination, Heart rate at rest, blood pressure, maximum load level, VE/VCO2, PetCO2, VE/VCO2 slope, VO2, Respiratory rate, VD/VT, SpO2, RER, Borg score, FEV1, FVC
Valve opening and closure behavior | Up to 5 Years Follow-Up
  Measurement tool: Echocardiography + Magnetic resonance imaging Parameter: 1.) blood flow velocity / stenosis, 2.) stiff leaflet, 3.) valve opening area Decision rule: blood flow velocity >4 m/s, abnormal or no leaflet motion when compared to neighboring leaflets, > 0.70 for 17 diameter, > 0.85 for 19, > 1.05 for 21, > 1.25 for 23, > 1.45 for 25, > 1.70 for 27, 1.95 for 29, and 2.25 for 31 mm annulus diameter
Valve closure behavior | Up to 5 Years Follow-Up
  Measurement tool: Echocardiography + Magnetic resonance imaging Parameter: 1.) vena contracta, 2.) Proximal Isovelocity Surface Area (PISA) radius, 3.) Effective regurgitation orifice area (EROA=2π*r2*Va/Vmax), (iv) sagging leaflet Decision rule: 1.) less than or equal to 15% of the diameter of PA/stent at a Nyquist limit of 0.5-0.6 m/s, frame rate >20/sec, gain adjusted, sector small, 2.) equal or minor to 4 mm at a Nyquist limit of 0.2-0.4 m/s, frame rate >20/sec, gain adjusted, variance off, sector small, 3.) < or equal to 3% of the total cross-sectional area of the valve, 4.) n.a
Heart rhythm | Up to 5 Years Follow-Up
  Assessment if new or higher grade of cardiac arrhythmia occured, i.e. newly ventricular extra systoly
Position and condition of the stent and structures | Up to 1 Year Follow-Up
  Measurement tool: Echocardiography + Magnetic resonance imaging + computed tomography Parameter: 1.) GrOwnValve annulus, 2.) no broken struts of the valve stent Decision rule: 1.) +/- 1.5 mm from the native pulmonary valve annulus, 2.) n.a.
Blood flow | Up to 1 Year Follow-Up
  Assessment of backflow and volume of blood by echo + MRI

SECONDARY OUTCOMES:
Availability of pericardium or other tissue for preparation of autologous pulmonary valve graft | Procedure (intra-operatively)
  Visual assessment of pericardium
Post-procedure length of stay | Up to day of discharge ( ≤ 30 days)
  Post-procedure hospital stay in days.
Ventilation time | Procedure (intra-operatively)
  Timepoints: Procedure Assessment: How long was the ventilation time for each patient within the allocation?
Freedom from conduction disturbances and arrhythmias need for permanent pacemaker implantation | Up to 3 months Follow-Up
  Timepoints: Procedure + Discharge + Visit 1 Assessment: Is the implantation of a permanent pacemaker necessary due to disturbances or arrhythmias?
(Re-)Hospitalization | Up to 60 months (5 years) Follow-Up
  Timepoints: Discharge, Visit 1, Visit 2, Visit 3, Visit 4, Visit 5, Visit 6, Visit 7, Visit 8 Assessment: Is a (Re-)Hospitalization necessary due to procedure- or device-related complications?
Comparison of pericardiectomy (if applicable) via thoracoscopy vs. thoracotomy | Procedure (intra-operatively)
  Timepoints: Procedure Assessment: How was the pericardiectomy conducted, via thoracoscopy or thoracotomy
Procedure-related death, major bleeding, reoperation, and other complications. | Follow-Up for 6 months
  Assessment of the GrOwnValve procedure's safety. Therefore, procedure-related death, major bleeding, reoperation, and other complications will be documented combined and individually for 6 months. Whenever the procedure evaluates as "not safe", the reasons will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Schmitt, Dr., Study Director — Charité UNiveristätsmedizin Berlin, Deutsches Herzzentreum der Charité
Locations (1):
- Charité Universitätsmedizin Berlin, Campus Virchow Klinikum, Deutsches Herzzentrum der Charité, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No